CLINICAL TRIAL: NCT01150734
Title: Transcranial Direct Current Stimulation (tDCS)-Boosted Changes in Muscle Evoked Potentials (MEP) in Depressed and Schizophrenic Patients Reveal Deficits in Neuromodulation
Brief Title: Neuromodulation in Depressed and Schizophrenic Patients - Changing MEP (Muscle Evoked Potentials) by tDCS (Transcranial Direct Current Stimulation)
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Palm, U, MD, Dept. of Psychiatry and Psychotherapy
Other Study IDs: 07/2009
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Schizophrenia; Depression
Keywords: differences of Muscle evoked potentials (MEP) in psychiatric illnesses; differences in neuromodulation; normalization of neuromodulation after pharmacological treatment
MeSH Terms: conditions — Schizophrenia; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Muscle evoked potentials (MEP) are supposed to different in schizophrenic and depressed patients, compared to a sample of healthy volunteers. Transcranial Magnetic Stimulation (TMS)-evoked MEP are measured in all three groups at baseline and after tDCS (2 mA, 20 minutes). MEP amplitudes are supposed to normalize quickly in healthy volunteers, to stay diminished in depressed patients and to stay elevated in schizophrenic patients. These differences should disappear after regular pharmacological treatment. Outcome measures will be done in week 2 and week 4.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be in the condition to understand the patient-information, as well as the necessary examinations.
* He/she must be able to give a written consent.
* No medication at least three weeks before enrollment.

Exclusion Criteria:

* Existence of a care/legal incapacity
* Existing pregnancy
* Severe psychiatric illness (with exception of affective disorder)
* Acute suicidality
* Drug-, medication- or alcohol dependence
* Dementia according to DSM IV / ICD 10-criterions
* Severe brain infarctus in the anamnesis
* Indications of structural damage of the basal ganglia or the brain stem
* Severe neurological disorders (e.g. M. Parkinson, epilepsy, discus-prolapse, dementia, systemic neurological illnesses, normal pressure hydrocephalus, cerebrovascular diseases, elevated intracranial pressure, in the last 6 months, polyneuropathies).
* Severe other medical conditions, like manifest arterial hypertonia, severe heart disease, pacemakers, respiratory failure, malignant illnesses all type, also in the history, active infectious diseases, skeletal disorders (like M. Paget, osteoporosis with spontaneous fractures, fresh fractures) Other circumstances, that speaks against a participation of the patient pinion of Medical Doctor at this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 depressed patients 15 schizophrenic patients 15 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Decreased MEP amplitudes in depressed patients | at baseline
  MEP amplitudes are supposed to be lower than in healthy controls or schizophrenic patients

SECONDARY OUTCOMES:
Elevated MEP amplitudes in schizophrenic patients | at baseline
  MEP amplitued are supposed to be elevated in schizophrenic patients in comparison to depressed patients or healthy controls
Normalization of MEP amplitudes after drug treatment | 4 weeks after baseline
  MEP aplitued of schizophrenic patients are supposed to normalize after regular drug treatment within 4 weeks.
Normalization of MEP amplitudes after drug treatment | 4 weeks after baseline
  MEP aplitued of depressed patients are supposed to normalize after regular drug treatment within 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Padberg, MD, Study Director — Ludwig-Maximilian-University
Locations (1):
- Ludwig-Maximilians-University, Munich, Germany

REFERENCES:
- See also: Related Info — http://psywifo.klinikum.uni-muenchen.de/forschung/tms/index.html